CLINICAL TRIAL: NCT05117372
Title: ANALYSIS OF INFLAMMATORY REACTIONS OBSERVED IN BRONCHOALVEOLAR LAVAGES (BALS) PERFORMED FOR INFILTRATIVE LUNG DISEASE THAT COMPLICATE ANTI PD-(L)1 IMMUNOTHERAPIES
Brief Title: ANALYSIS OF INFLAMMATORY REACTIONS OBSERVED IN BRONCHOALVEOLAR LAVAGES (BALS)
Acronym: LBA-PI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-A01626-33
Record Dates: First submitted 2021-08-06; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-08

CONDITIONS: Lung Cancer
Keywords: anti PD-(L)1; Diffuse infiltrative lung disease
MeSH Terms: conditions — Lung Neoplasms | interventions — Therapeutics; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients treated with with immunotherapy and developing diffuse infiltrative lung disease (Active Comparator): Group 1: Patients treated for cancer with immunotherapy and developing diffuse infiltrative lung disease
  Interventions: Other: treatment with immunotherapy and diffuse infiltrative lung disease
- Patients not treated with immunotherapy and requiring carcinologic lobectomy (Placebo Comparator): Group 2: Patients with lung cancer not treated with immunotherapy and requiring carcinologic lobectomy
  Interventions: Other: Patients requiring carcinologic lobectomy

INTERVENTIONS:
Other: treatment with immunotherapy and diffuse infiltrative lung disease — Patients treated with with immunotherapy and developing diffuse infiltrative lung disease
  Arms: Patients treated with with immunotherapy and developing diffuse infiltrative lung disease
Other: Patients requiring carcinologic lobectomy — Patients requiring carcinologic lobectomy
  Arms: Patients not treated with immunotherapy and requiring carcinologic lobectomy

SUMMARY:
Immunological toxicities associated with immune checkpoint inhibitor (ICI) monoclonal antibodies are unpredictable autoimmune and inflammatory pathologies that can affect all treated patients. Some of these events are severe and occur in 15-20% of patients treated with Programmed Death 1 (PD-1) antibodies.

The study of cellular immunological characteristics within tissues affected by toxicities and the interactions between the different actors of these toxicities aims at improving the knowledge concerning the mechanisms of these toxicities, but also at being able to specify the unexpected effects of ICIs on cells of the immune system, outside the tumor microenvironment.

Diffuse infiltrative lung disease is one of the most frequent and severe toxicities encountered in patients treated with anti PD-(L)1; either for bronchial cancer, melanoma or any other type of cancer. Patients developing this type of complication benefit from cytological, bacteriological, mycological and molecular analyses of intra-alveolar constituents obtained by bronchoalveolar lavage (BAL) performed during bronchial fibroscopy as part of their routine care. These analyses help to confirm the diagnosis of alveolitis, to specify the cellular characteristics of alveolar inflammation and to eliminate differential diagnoses of ICI toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject (≥ 18 years old)
* Patient having consented to the research

Group 1:

* Patient with cancer who was treated with immunotherapy
* Appearance of CT lung abnormalities during immunotherapy, not related to cancer
* With high suspicion of infiltrative lung disease:
* Pneumopathy (CTCAE version 5 classification).
* Patients requiring bronchial fibroscopy with BAL

Groups 2:

* Patient with lung cancer with peripheral tumor
* Requires surgical pulmonary lobectomy in the operating room

Exclusion Criteria:

* Patient treated or having been treated in the last 2 months with corticosteroid therapy
* Patient treated with immunosuppressant and/or cyclophosphamide, and/or Anti-TNF α in the last 12 months
* Absence of consent
* Patient under curatorship, guardianship or safeguard of justice
* Pregnant woman
* Group 1:
* Patient with respiratory failure

Groups 2:

* Patient with lung cancer with proximal or endobronchial tumor
* Patients requiring bilobectomy or pneumonectomy
* Patient who has been treated with immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-08-17 (Estimated); Study Completion 2024-02-17 (Estimated)

PRIMARY OUTCOMES:
Expression levels of cellular and soluble actors involved in the occurrence of pulmonary toxicities associated with antitumor immunotherapies | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson, France